CLINICAL TRIAL: NCT03998579
Title: The Effect of Physical Rehabilitation Among Patients Undergoing Radical Cystectomy Due to Urinary Bladder Cancer - the CanMoRe Study
Brief Title: Physical Rehabilitation Among Patients Undergoing Radical Cystectomy Due to Urinary Bladder Cancer
Acronym: CanMoRe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Hagströmer, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/2214-31/4
Record Dates: First submitted 2019-06-07; First posted 2019-06-26 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized exercise (Experimental): The intervention group get a referral to physiotherapist in Primary Health Care in Stockholm County Council, close to where they live. Within the third week after discharge, the patients begin twelve weeks of biweekly exercise. The physical exercise is individually targeted aerobic and strength exercises, based on international recommendations for persons with cancer disease. The program is approved by resposible surgeons.
  Interventions: Other: The CanMoRe programme
- Active control group (Active Comparator): Oral and written information of a home-based exercise programme and information of supportive techniques to improve physical activity
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: The CanMoRe programme — An exercise intervention in Primary Health Care
  Arms: Individualized exercise
Other: Home exercise — An active control group
  Arms: Active control group

SUMMARY:
The main objective of the CanMoRe study is to evaluate the impact of a standardized and individually adapted exercise intervention in Primary Health Care aiming at improving physical function (primary outcome) and habitual physical activity, health related quality of life, fatigue and psychological well-being in patients undergoing radical cystectomy due to urinary bladder cancer.

DETAILED DESCRIPTION:
The most common treatment for solid cancer tumours is surgery, often in combination with chemo- and/or radiotherapy. To minimise the postoperative complications is important in today's health care. Early mobilisation at the ward and physical activity at home after discharge, have been shown to be important parts to reduce complications. Common complications after abdominal surgery are postoperative pulmonary complications and venous thrombosis. One of the conditions that suffers the most from different kinds of postoperative complications is radical cystectomy due to urinary bladder cancer. Complications after radical cystectomy could be direct related to the patients' high age and also high degree of comorbidity.

There is today strong evidence that physical activity has a positive impact on health, survival and quality of life. Patients who have been treated for urinary bladder cancer are not sufficiently physical active and suffer from readmissions to hospital due to complications. Therefore, there is a need for developing and testing a physical rehabilitation programme to support patients who have a radical cystectomy, in the early postoperative period.

The CanMoRe study is a randomized controlled trial with a single-blinded design evaluating an exercise intervention in Primary Health Care as part of the CanMoRe programme. In addition, a qualitative study (interviews) on patient's experience of the programme will be conducted as well as data gathered on factors that might influence the implementation of the programme.

Then CanMoRe programme consists of preoperative information, the Activity Board used for enhanced mobilization during hospital stay, a 12-week, (1 h, 2 times/week) standardized and individually adapted exercise intervention in Primary Health Care and behavioral support for daily physical activity. The CanMoRe programme is evaluated in two steps, i.e. the in-hospital intervention using the Activity Board (published) and the exercise intervention in Primary Health Care reported herein.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for a robotic assisted laparoscopic radical cystectomy due to urinary bladder cancer at the Karolinska University Hospital Solna will be included in the trial. The patients should be able to talk and understand Swedish, live in the Stockholm County Council area and be mobile with or without walking aid.

Exclusion Criteria:

* Patients who will undergo radical cystectomy on a non-curative basis will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test | Change from baseline to after 12 weeks intervention
  The test reproduces activity of daily living at a sub maximal level. Output: meters Score: 0-900.

SECONDARY OUTCOMES:
ActivPAL accelerometer | Measurement 1: Baseline, Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge
  Habitual physical activity, measured for 7 consecutive days. Output: number of steps per day.
Chair stand test | Measurement 1: Baseline, Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge
  Measure of leg strength. Output: Scale 0-30
Hand grip strength | Measurement 1: Baseline, Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge,
  Measure of hand grip strength (Jamar hand dynamometer). Output: Kilo 0-60
European Organisation for Research and Treatment of Cancer (EORTC) Quality of life for cancer patients QLQ-C30 | Measurement 1: Baseline Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge
  Health related quality of life. Output: Scale 0-100. A higher score is worse outcome. For more information see https://qol.eortc.org/questionnaires/
EORTC QLQ-BLM30 | Measurement 1: Baseline Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge
  Health related quality of life specific for bladder cancer Output: Scale 0-100, a higher score is worse
Piper Fatigue Scale | Measurement 1: Baseline, Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge
  Fatigue. Output: Scale 0-10. A higher score is worse, i.e more fatigue
Numeric rating scale (NRS) | Measurement 1: Baseline, Measurement 2: After 12 weeks intervention. Measurement 3: 1 year after discharge
  Pain. Output: Scale 0-10, A higher score is worse i.e more pain
Hospital Anxiety and Depression Scale (HADS) | Measurement 1: Baseline, Measurement 2: 12 weeks. Measurement 3: 1 year after discharge
  Psychological wellbeing. Output: Scale 0-21. A higher score is worse
Readmission | Collected from journals using standardized time frames at 30 and 90 days
  Readmissions to hospital. Output: Yes/No
Complications | Collected from journals using standardized time frames at 30 and 90 days
  Complications such as Pneumonia Output: according to Clavien - Dindo classification
Six-minute walk test | Measurement 3: 1 year after discharge
  The test reproduces activity of daily living at a sub maximal level. Output: meters Score: 0-900.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hagstromer, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porserud A, Karlsson P, Rydwik E, Aly M, Henningsohn L, Nygren-Bonnier M, Hagstromer M. The CanMoRe trial - evaluating the effects of an exercise intervention after robotic-assisted radical cystectomy for urinary bladder cancer: the study protocol of a randomised controlled trial. BMC Cancer. 2020 Aug 26;20(1):805. doi: 10.1186/s12885-020-07140-5. PMID 32842975
- [Derived] Porserud A, Aly M, Steinertz H, Rydwik E, Hagstromer M. Exercise in primary care after robot-assisted radical cystectomy for urinary bladder cancer - effects on postoperative complications: a secondary analysis of a randomised controlled trial. Scand J Urol. 2024 Dec 18;59:193-199. doi: 10.2340/sju.v59.42589. PMID 39692276
- [Derived] Porserud A, Karlsson P, Aly M, Rydwik E, Torikka S, Henningsohn L, Nygren-Bonnier M, Hagstromer M. Effects of an exercise intervention in primary care after robot-assisted radical cystectomy for urinary bladder cancer: a randomised controlled trial. BMC Cancer. 2024 Jul 24;24(1):891. doi: 10.1186/s12885-024-12647-2. PMID 39048933
- See also: The link to the larger project to which this RCT belong — https://ki.se/en/nvs/the-abdmore-project-2016-2020